CLINICAL TRIAL: NCT01898247
Title: Use of Simulation-Based Mastery Learning for Resident Thoracentesis Training to Improve Patient Outcomes
Brief Title: Use of Simulation-Based Mastery Learning for Thoracentesis to Improve Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jeffrey Barsuk, Associate Professor of Medicine, Northwestern University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Other
Other Study IDs: STU00069024
Record Dates: First submitted 2013-07-05; First posted 2013-07-12 (Estimated); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: Misadventure During Thoracentesis
Keywords: Thoracentesis; Simulation Based Mastery Learning; Medical Education; Length of Stay; Cost of Care

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Traditionally-trained Procedures (No Intervention): Patients who undergo thoracentesis procedures by traditionally-trained residents who have not undergone simulation-based mastery learning.
- Simulator-trained Procedures (Experimental): Patients who undergo thoracentesis procedures by residents who have undergone simulation-based mastery learning.
  Interventions: Other: Simulation-based mastery learning

INTERVENTIONS:
Other: Simulation-based mastery learning — Internal Medicine residents are randomly selected to undergo simulation-based mastery learning.
  Arms: Simulator-trained Procedures

SUMMARY:
The goal of the proposed research is to investigate the use a medical simulation and mastery learning (where all learners must reach a high standard before completion of training) curriculum to improve internal medicine residents' skills when performing thoracentesis procedures (remove fluid from around the lung) on patients. Additionally, we will evaluate how these skills affect patient outcomes by comparing thoracenteses performed by simulator-trained residents to those who have "traditional" training. This project will evaluate these overall hypotheses: simulation-based training using the mastery learning approach improves medicine resident's thoracentesis skills and improves patient outcomes and satisfaction.

DETAILED DESCRIPTION:
Given medical procedures are the second most common cause of the complications that afflict 3% of hospitalized patients, simulation-based mastery learning should be applied to procedures done in all medical centers. In academic hospitals, bedside procedures such as thoracentesis procedures are often performed by unsupervised medical trainees. Traditionally, medical trainees learn procedures relying on the historic "see one, do one, teach one" mentality. Unfortunately, this approach subjects patients to procedures before trainees are competent.

Through the use of medical simulation, medical educators can increase the essential knowledge and skills of trainees while assuring procedural competence and reducing patient exposure to undue risk. Medical simulation training using the mastery learning model improves clinical skills and reduces the risk of procedure-associated injury. Our research group pioneered the use of this evidence-based approach for teaching medical trainees. Mastery learning requires that all trainees demonstrate a uniformly high level of skill before training completion. This ensures competence on a medical simulator before actual patient encounters.

ELIGIBILITY:
Inclusion Criteria:

* Patients:

  * undergoing a thoracentesis procedure
  * on internal medicine or hospitalist ward service
  * English or Spanish Speaking
* 2nd and 3rd year internal medicine residents

Exclusion Criteria:

* Cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2012-12; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Simulation based mastery learning for resident thoracentesis training will increase patient satisfaction and safety. | 30 months
  Thoracentesis skills will be measured using a checklist on the simulator and on actual patients during direct observations. Satisfaction with procedures done by a referred service or at the bedside by simulator-trained residents will be measured by patient reported confidence levels in procedure performer, perception of delay, and comfort during the procedure. Patient safety will be measured by assessing documented complication rates such as: pneumothorax, bleeding, infection, reexpansion pulmonary edema, and significant pain. Additionally, length of stay and hospital costs will be compared between patients undergoing thoracentesis by simulator-trained residents versus referred services (or traditionally-trained residents).

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey H. Barsuk, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Derived] Barsuk JH, Cohen ER, Williams MV, Scher J, Feinglass J, McGaghie WC, O'Hara K, Wayne DB. The effect of simulation-based mastery learning on thoracentesis referral patterns. J Hosp Med. 2016 Nov;11(11):792-795. doi: 10.1002/jhm.2623. Epub 2016 Jun 8. PMID 27273066